CLINICAL TRIAL: NCT04803864
Title: A Randomized Controlled Trial to Evaluate the Safety and Efficacy of Roxadustat in Patients With Acute ST Elevation Myocardial Infarction
Brief Title: Study of Roxadustat in the Treatment of Acute Myocardial Infarction
Acronym: ROXAMI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, RUIYAN ZHANG, Director of Cardiology Department, Chief Physician, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHDC2020CR2023B
Record Dates: First submitted 2021-02-02; First posted 2021-03-18 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST Elevation Myocardial Infarction; Roxadustat; Infarct Size; Cardiac MRI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — roxadustat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roxadustat (Experimental): Early and short-term Roxadustat treatment
  Interventions: Drug: Roxadustat
- Control (No Intervention): Patients only receive conventional therapies as recommended by guidelines.

INTERVENTIONS:
Drug: Roxadustat — Orally 100mg, 3 times per week for 2 weeks First dose administered immediately after successful PCI.
  Other Names: Evrenzo
  Arms: Roxadustat

SUMMARY:
Depite successful primary percutaneous coronary intervention (PCI) and standardized medical treatment, prognosis of acute ST-elevation myocardial infarction patents are still a poor, with high morality and various complications such as heart failure. Roxadustat is a new drug targeting hypoxia-inducible factor prolyl hydroxylase (HIF-PH) inhibition and has shown promising effect in reducing infarct size in pre-clinical studies.

This study aims to evaluate the efficacy and safety of early and short-term administration of roxadustat in the treatment of acute ST-elevation myocardial infarction.

DETAILED DESCRIPTION:
This study is an open-label, paralleled, randomized controlled trial. It aims to evaluate the efficacy and safety of early and short-term administration of roxadustat in the treatment of acute ST-elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Acute STEMI (ST segment elevation myocardial infarction) diagnosed by ST elevation
* Coronary angiography within 12 hours of symptom onset, with TIMI flow grade 0 - 1 of culprit vessel
* Primary PCI with TIMI flow grade 2 - 3 after successful intervention
* Capable and willing to provide informed consent and capable of completing study visits

Exclusion Criteria:

* Previous acute myocardial infarction history
* Cardiogenic Shock at admission
* Previously treated by roxadustat
* Contraindications of roxadustat treatment
* Contraindication of Cardiac MRI (e.g. eGFR < 30 ml/min, pacemaker, metal prosthesis, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Infarct Size | 30 days
  Infarct size as a percentage of LV mass measured on delayed-enhanced CMR imaging 30 days post-MI compared to control

SECONDARY OUTCOMES:
MACE | 0 - 1 year
  Major adverse cardiovascular events (MACE) within 1 year follow-up.
Left Ventricular Function | 1 month, 6 months, 1 year
  Left ventricular end diastolic volume (LVEDV), Left ventricular end systolic volume (LVESV), Left ventricular ejection fraction (LVEF) changes during 1 year follow-up
Cardiac enzymes - peak concentration | 0 - 3 days
  Peak Plasma Concentration (Cmax) of CK-MB, TnI and CK
Cardiac enzymes - Area under curve | 0 - 3 days
  Area under the plasma concentration versus time curve (AUC) of CK-MB, TnI and CK

OTHER OUTCOMES:
Myocardial fibrosis | 30 days
  Fibroblast activation protein inhibitor (FAPI) tracer uptake in myocardium if selected patient underwent spontaneous PET/MR scan

CONTACTS AND LOCATIONS:
Overall Officials: Ruiyan Zhang, M.D., Ph.D., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data by contacting principle investigator of this study. Requests for IPD will be recieved, but this does not mean all requests will be shared by the investigators.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after the end of this study
Access Criteria: Please contact the investigators through email in the time frame.

REFERENCES:
- [Background] Howell NJ, Tennant DA. The role of HIFs in ischemia-reperfusion injury. Hypoxia (Auckl). 2014 Jul 30;2:107-115. doi: 10.2147/HP.S49720. eCollection 2014. PMID 27774470
- [Background] Sousa Fialho MDL, Abd Jamil AH, Stannard GA, Heather LC. Hypoxia-inducible factor 1 signalling, metabolism and its therapeutic potential in cardiovascular disease. Biochim Biophys Acta Mol Basis Dis. 2019 Apr 1;1865(4):831-843. doi: 10.1016/j.bbadis.2018.09.024. Epub 2018 Sep 25. PMID 30266651
- [Background] Schreiber T, Salhofer L, Quinting T, Fandrey J. Things get broken: the hypoxia-inducible factor prolyl hydroxylases in ischemic heart disease. Basic Res Cardiol. 2019 Mar 11;114(3):16. doi: 10.1007/s00395-019-0725-2. PMID 30859331
- [Background] Chen N, Hao C, Peng X, Lin H, Yin A, Hao L, Tao Y, Liang X, Liu Z, Xing C, Chen J, Luo L, Zuo L, Liao Y, Liu BC, Leong R, Wang C, Liu C, Neff T, Szczech L, Yu KP. Roxadustat for Anemia in Patients with Kidney Disease Not Receiving Dialysis. N Engl J Med. 2019 Sep 12;381(11):1001-1010. doi: 10.1056/NEJMoa1813599. Epub 2019 Jul 24. PMID 31340089
- [Background] Deguchi H, Ikeda M, Ide T, Tadokoro T, Ikeda S, Okabe K, Ishikita A, Saku K, Matsushima S, Tsutsui H. Roxadustat Markedly Reduces Myocardial Ischemia Reperfusion Injury in Mice. Circ J. 2020 May 25;84(6):1028-1033. doi: 10.1253/circj.CJ-19-1039. Epub 2020 Mar 24. PMID 32213720
- [Background] Groenendaal-van de Meent D, den Adel M, Rijnders S, Krebs-Brown A, Kerbusch V, Golor G, Schaddelee M. The Hypoxia-inducible Factor Prolyl-Hydroxylase Inhibitor Roxadustat (FG-4592) and Warfarin in Healthy Volunteers: A Pharmacokinetic and Pharmacodynamic Drug-Drug Interaction Study. Clin Ther. 2016 Apr;38(4):918-28. doi: 10.1016/j.clinthera.2016.02.010. Epub 2016 Mar 4. PMID 26947173